CLINICAL TRIAL: NCT06873451
Title: 3D Comparison Effects of Two Different Surgical Timings in Orthognathic Surgery on Root Resorption and Soft Tissues: Surgery First vs. Surgery Early
Brief Title: Effects of Orthognathic Surgery on Root Resorption and Soft Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gokhan Coban (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Gokhan Coban, ASSOC. PROF. DR., TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-655
Record Dates: First submitted 2025-02-13; First posted 2025-03-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Orthodontics; Orthognathic Surgical Procedures
Keywords: Orthognathic surgery; Surgery first; surgery early; dehiscence; Fenestration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery First (Experimental): Patients in this group started with surgical treatment directly without receiving orthodontic treatment and started orthodontic treatment after surgery.
  Interventions: Procedure: Surgery First
- Surgery Early (Experimental): Patients in this group were referred to orthognathic surgery after receiving orthodontic treatment for an average of 6-8 months, and their orthodontic treatments continued after surgery.
  Interventions: Procedure: Surgery Early

INTERVENTIONS:
Procedure: Surgery First — One month after surgery, patients were called for an appointment and lower and upper brackets were placed. Treatment was completed when right-left Class I canine and molar relationships and ideal overjet and overbite relationships were achieved.
  Arms: Surgery First
Procedure: Surgery Early — The patients were directed to surgery with the upper and lower bonds applied at their first appointment and the brackets in their mouths. After surgery, treatment continued until the right-left Class I canine and molar relationship and the ideal overjet and overbite relationship were achieved.
  Arms: Surgery Early

SUMMARY:
The aim of this study is to evaluate the three-dimensional tomographic and photographic evaluation of the provision of two different orthognathic surgeries on hard and soft tissues with informative Class III deformity due to maxillary retrognathia and mandibular prognathia.

DETAILED DESCRIPTION:
Patients who will undergo non-extraction surgery will be randomized as 'Pre-Surgery' (SEC) and 'Early Surgery' (EC). Maxillary advancement and mandibular recession will be calculated and a total of 24 patients, 12 in each group, will be included in the study. Millimetric (length, dehiscence, fenestration) and volumetric measurements and soft tissue anthropometric points will be measured in three-dimensional recordings taken at the beginning of treatment (T0) and after debonding (T1). Cone beam computed tomography (CBCT) images will be transferred to NNT and 'Mimics 18.0' programs for measurements. Three-dimensional photographs will be evaluated in the 3dMDvultus program. Shapiro-Wilk test will be used for normality, 'two independent samples t-test' and 'Mann Whitney U test' will be used for intra-group and inter-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* They must be over 18 years of age,
* Skeletal Class III malocclusion and need double jaw orthognathic surgery,
* Minimum crowding (patients with crowding between 0-3 mm),
* Complete 3D records before surgery and at the end of treatment,
* No decay on their teeth,
* Good oral hygiene,
* Healthy periodontal tissues.

Exclusion Criteria:

* History of trauma,
* Congenital anomalies or craniofacial deformities
* Congenital tooth loss (excluding wisdom teeth)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Tooth length measurement (mm) | up to 15 months
  Root length of maxillary incisors will be measured using cone-beam computed tomography (CBCT). Data will be reported as mean change (± SD).
Tooth volume measurement (mm^3) | up to 15 months
  Root volume of maxillary incisors will be measured using cone-beam computed tomography (CBCT). Data will be reported as mean change (± SD).

SECONDARY OUTCOMES:
Soft tissue measurement (3D) | up to 15 months
  Three-dimensional stereophotogrammetry will be used to assess changes in facial soft tissue profile, including convexity and lip-chin relationships. Results will be summarized as mean changes (± SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry Department of Orthodontics, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juggins KJ, Nixon F, Cunningham SJ. Patient- and clinician-perceived need for orthognathic surgery. Am J Orthod Dentofacial Orthop. 2005 Dec;128(6):697-702. doi: 10.1016/j.ajodo.2004.09.022. PMID 16360908
- [Background] Hernandez-Alfaro F, Guijarro-Martinez R. On a definition of the appropriate timing for surgical intervention in orthognathic surgery. Int J Oral Maxillofac Surg. 2014 Jul;43(7):846-55. doi: 10.1016/j.ijom.2014.02.007. Epub 2014 Mar 13. PMID 24631424
- [Background] Millesi GA, Zimmermann M, Eltz M. Surgery First and Surgery Early Treatment Approach in Orthognathic Surgery. Oral Maxillofac Surg Clin North Am. 2023 Feb;35(1):71-82. doi: 10.1016/j.coms.2022.06.010. Epub 2022 Nov 3. PMID 36336597
- [Background] Hernandez-Alfaro F, Guijarro-Martinez R, Molina-Coral A, Badia-Escriche C. "Surgery first" in bimaxillary orthognathic surgery. J Oral Maxillofac Surg. 2011 Jun;69(6):e201-7. doi: 10.1016/j.joms.2011.01.010. Epub 2011 Apr 5. No abstract available. PMID 21470740